CLINICAL TRIAL: NCT02727556
Title: Physiological Response and Visual Attention to Visual Food Images in Healthy Subjects and in Functional Dyspepsia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Inseon Lee, MS, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 041/2016BO2
Record Dates: First submitted 2016-03-21; First posted 2016-04-04 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Functional Dyspepsia
Keywords: skin conductance response; facial muscle activity; heart rate variability; eyetracking

ARMS (2):
- Functional dyspepsia patient (Experimental): Visual stimuli of food and non-food images will be presented to patients. Non-food images include positive, neutral, negative emotional pictures.
  Interventions: Behavioral: visual images
- Healthy (Experimental): Visual stimuli of food and non-food images will be presented to participants. Non-food images include positive, neutral, negative emotional pictures.
  Interventions: Behavioral: visual images

INTERVENTIONS:
Behavioral: visual images

SUMMARY:
In functional dyspepsia (FD), abnormal cognitive and emotional changes such increased sensitization, anxiety, and depression scores have been reported in addition to the peripheral changes in gastrointestinal tract functions. In this study, investigators will evaluate the activity of autonomic nervous system, emotional response, and visual attention to food and non-food images in 30 male and female FD patients and 30 age/gender-matched healthy volunteers. These data will provide a new finding of the influence of impaired cognitive processing of food on symptom generation in functional gastrointestinal disorder patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, volunteering adults BMI: 18-25 kg/m² right-handed Age: 18-65 years Capacity to give informed consent For FD patients, Diagnosis of functional dyspepsia over the last 12 months certified by a medical record Inconspicuous gastroscopy during the last 6 months certified by a medical record

Exclusion Criteria:

* Visual impairment Severe psychiatric illness (e.g. schizophrenia, severe depression (BDI-II:29-63)), substance dependence and abuse Intake of antidepressants / antipsychotics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Psychological response | 1-2 years
  Skin conductance response
Psychological response | 1-2 years
  heart rate variability
Psychological response | 1-2 years
  facial muscle contraction
visual attention | 1-2 years
  eyemovement

SECONDARY OUTCOMES:
Subjective rating | 1-2 years
  fullness (visual analog scale)
Subjective rating | 1-2 years
  satiation (visual analog scale)
Subjective rating | 1-2 years
  nausea (visual analog scale)
Subjective rating | 1-2 years
  pain (visual analog scale)
Subjective rating | 1-2 years
  mood (visual analog scale)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Enck, Prof, Principal Investigator — Psychosomatic Medicine and Psychotherapy Department, University of Tübingen, Tübingen, Germany
Locations (1):
- Psychosomatic Medicine and Psychotherapy Department, University of Tübingen, Tübingen, Germany, Tübingen, Germany